CLINICAL TRIAL: NCT06799221
Title: Expanded Access Program (EAP) for Obecabtagene Autoleucel (obe-cel) Out-of-specification (OOS) in Adult Patients with Acute Lymphoblastic Leukemia
Brief Title: Expanded Access Program for OOS Obe-cel
Status: Available | Type: Expanded Access
Sponsor: Autolus Limited (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: AUTO1-OS1
Record Dates: First submitted 2025-01-23; First posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Lymphoblastic Leukemia, Acute, Adult; B Cell ALL
Keywords: Relapsed B cell acute lymphoblastic leukemia; Refractory B cell acute lymphoblastic leukemia; Adult acute lymphoblastic leukemia; Obecabtagene autoleucel (obe-cel); Obe-cel
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Biological: Out-of-specification obecabtagene autoleucel — Out-of-specification (OOS) obecabtagene autoleucel (obe-cel) given as a split-dose infusion based on tumor burden assessment at lymphodepletion according to the United States prescribing information.
  Other Names: OOS Obe-cel

SUMMARY:
The purpose of this program is to provide access to obe-cel treatment for adult patients with ALL who have undergone leukapheresis and had obe-cel manufactured from their blood cells but the product is deemed OOS (does not meet the specifications to be used commercially). The target patients for this study have limited options for treatment and repeat blood sampling is not feasible. The main aims of this study are (1) to provide adult patients with ALL with access to obe-cel and (2) to describe the safety profile of obe-cel (including CRS, ICANS, serious infections, secondary cancers, and any side effects) within the first 45 days after infusion of OOS obe-cel.

This study is a single-arm, open-label, multicenter expanded access program (EAP). The patient population included in this EAP will be adult patients diagnosed with recurring or refractory ALL who were prescribed obe-cel as part of their standard of care and are eligible for use under the approved local prescribing information.

To be in the study, patients must provide informed consent, be at least 18 years of age, have a confirmed diagnosis of ALL, be medically fit and stable to receive obe-cel, have had commercial obe-cel prescribed by their treating physician as per standard of care, and for whom remanufacturing is not clinically appropriate.

Patients cannot be in the study if they have a history of severe immediate allergic reaction to any drugs or metabolites of similar chemical classes as obe-cel, are a pregnant woman, or are receiving treatment in another study.

All data will be collected from information routinely recorded in the medical record. There is no formal hypothesis testing. Data will be analyzed descriptively (numbers, percentages and ranges, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patient (or legally authorized representative) is willing to provide informed consent.
* Patient must be 18 years of age or older.
* Patient must have a confirmed diagnosis of relapsed/refractory B cell ALL.
* Commercial obe-cel was indicated to the patient by their treating physician as per standard of care prior to leukapheresis.
* The final manufactured obe-cel does not meet the commercial release specifications.
* The final manufactured obe-cel is acceptable per joint assessment by Autolus and physician taking into account Autolus' release criteria.
* Remanufacturing (i.e., repeat leukapheresis and manufacturing) is not clinically appropriate per the treating physician's assessment.
* Patient deemed medically fit and stable to receive obe-cel infusions per their treating physician's evaluation.
* For females of childbearing potential (defined as < 24 months after last menstruation or not surgically sterile), a negative serum or urine pregnancy test must be documented at screening, prior to lymphodepletion therapy and confirmed before receiving the first dose of study treatment.
* For females who are not postmenopausal (< 24 months of amenorrhea) or who are not surgically sterile (absence of ovaries and/or uterus), 2 methods of contraception comprising 1 highly effective method of contraception together with a barrier method must be used during the treatment period and for at least 12 months after the last dose of study treatment. They must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the study and for 12 months after receiving the last dose of study drug.
* For males, it must be agreed that 2 acceptable methods of contraception are used (1 by the patient - usually a barrier method, and 1 highly effective method by the patient's partner) during the treatment period and for at least 12 months after the last dose of study treatment and that sperm will not be donated during the treatment period and for at least 12 months after the last dose of study treatment.

Exclusion Criteria:

* History of severe immediate hypersensitivity to any drugs or metabolites of similar chemical classes as obe-cel.
* Pregnant women.
* Active participation in an interventional trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Autolus Study Director, Study Director — Autolus Limited